CLINICAL TRIAL: NCT06526884
Title: Quasi-Randomized Evaluation of the UCLA Next Day Clinic (NDC)
Acronym: NDC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-000913
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Syncope; Congestive Heart Failure; Cellulitis; Pyelonephritis; AKI - Acute Kidney Injury; Diabetic Foot Infection; Osteomyelitis
Keywords: Patient safety; Cost effectiveness; Avoidable hospitalizations
MeSH Terms: conditions — Pneumonia; Syncope; Heart Failure; Cellulitis; Pyelonephritis; Acute Kidney Injury; Osteomyelitis

STUDY DESIGN:
Intervention Model Description: Randomized encouragement trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-initiated hospitalization (No Intervention): Patients with odd birthdays will be routed to standard-of-care ED-initiated hospitalization pathways.
- Next Day Clinic (Experimental): Patients with even birthdays who meet inclusion criteria will be given the option to receive care in the Next Day Clinic to avoid hospitalization.
  Interventions: Other: Next Day Clinic

INTERVENTIONS:
Other: Next Day Clinic — A dedicated Next Day Clinic team consisting of a clinician and nurse case manager will provide care and specialist referrals to patients within 24 hours of an ED visit that would have resulted in hospitalization without this novel hospital avoidance initiative.
  Arms: Next Day Clinic

SUMMARY:
The Next Day Clinic (NDC) is a quality improvement initiative that will be launched and operated by UCLA Health starting July 22, 2024. Its goals are to improve patient care and safety and to maximize cost effectiveness. The way it does this is by identifying patients in the ED who would normally be admitted for low-acuity conditions, and diverting them to a high-acuity clinic the following day called the NDC. This will help decompress the ED and the hospital, and allow for overall higher quality care. The Health System has partnered with UCLA's Healthcare Value Analytics and Solutions [UVAS] group which specializes in these types of program evaluations. The analysis conducted by the study team will be used to directly inform NDC operations, scaling, and future plans.

DETAILED DESCRIPTION:
NDC is a hospital avoidance model with the potential to simultaneously improve the quality and safety of acute care, reduce costs, and address hospital/ED overcrowding. This novel hospital avoidance program will divert patients from the ED who have been diagnosed with the following conditions and meet certain clinical criteria:

* Diabetic Foot Infection/Osteomyelitis
* Cellulitis
* Congestive Heart Failure
* Syncope
* Pyelonephritis/Urinary Tract Infection
* Pneumonia
* Acute Kidney Infection

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* About to be admitted through the ED for one of the NDC diagnoses or a synonym (per Study Protocol document), defined by the presence of a Plan to Admit order or Bed Request order, OR recently admitted under observation or inpatient status for one of the NDC diagnoses.
* Identified as at-risk for an avoidable hospitalization in the ED based on a pre-determined set of lab and vital parameters.
* Insurance that authorizes the patient to follow-up at UCLA Health, or self-pay
* Admitted or being admitted to an internal medicine service

Exclusion Criteria:

* Heart or lung transplant recipient with concern for graft dysfunction
* Pregnant
* Enrolled in hospice
* Admitted to a critical care service
* ED deems discharge unsafe due to complex social or medical factors
* Active malignant cancer (per Council of State and Territorial Epidemiologists value set)
* Pulmonary arterial hypertension (per Joint Commission value set)
* Undergoing workup for solid organ transplant
* Interstitial lung disease (including pulmonary fibrosis) (per Higher Level 7 value set)
* Requiring inpatient procedure or surgery defined by the presence of an anesthesia event or operating room encounter.
* The ED deems discharge unsafe due to complex social or medical factors.
* Transferred to an ineligible hospital

Note:

The Health System plans to limit the volume of referrals to the NDC by only referring patients who have an even birth date (this is more equitable than first-come-first-serve, because wage workers are more likely to come to the ED later in the day; even/odd birth date theoretically keeps more spots open for patients presenting to the ED later).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital (DAOH) | 30 days from index ED visit
  Cumulative number of days alive and not admitted or boarding in a hospital or emergency department

SECONDARY OUTCOMES:
Global health-related quality of life | 30 days from index ED visit
  Composite PROMIS-29+2 score (patient reported outcome measurement information system). PROMIS stands for Patient-Reported Outcomes Measurement Information System. High scores mean more of the concept being measured.
Patient experience | 30 days from index ED visit
  Measured by PSQ-18 (patient satisfaction questionnaire). PSQ stands for Patient Satisfaction Questionnaire. High scores indicate higher levels of satisfaction.
Financial analysis | Through study completion, an average of 12 months
  Total cost per day of treatment
Cost effectiveness analysis | Through study completion, an average of 12 months
  Total cost per day alive and out of hospital
Hospitalizations avoided | Through study completion, an average of 12 months
  Each NDC referral with a preceding Plan to Admit order or Bed Request order (regardless of treatment arm) will be considered an avoided hospitalization, given that the presence of one of these orders establishes that the counterfactual for NDC treatment in hospitalization.
Hospital bed-days saved | Through study completion, an average of 12 months
  For each referral to the NDC, the number of hospital bed-days saved will be established by using the mean length of stay for patients treated per-protocol in the control condition matched for the same presenting illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be uploaded to a data repository system such as Vivli.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT06526884/SAP_001.pdf